CLINICAL TRIAL: NCT03606187
Title: Stimgenics Open-Label, Post Market Study: A Clinical Trial to Study the Effects of Stimgenics Spinal Cord Stimulation (SGX-SCS) Programs in Treating Intractable Chronic Back Pain
Brief Title: Stimgenics Open-Label, Post Market Study
Acronym: SGX-SCS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stimgenics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGEN-2018PM2
Record Dates: First submitted 2018-07-12; First posted 2018-07-30 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Chronic Low Back Pain
Keywords: Back Pain, Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Arm (Experimental): Subjects randomized to this arm will receive test treatment
  Interventions: Device: Stimgenics SCS Programming Approach
- Control Arm (Active Comparator): Subjects randomized to this arm will receive control treatment
  Interventions: Device: Standard SCS Programming Approach

INTERVENTIONS:
Device: Stimgenics SCS Programming Approach — Stimgenics SCS Programming approach Using Intellis(TM) SCS system
  Arms: Test Arm
Device: Standard SCS Programming Approach — Standard SCS Programming approach using Intellis(TM) SCS system
  Arms: Control Arm

SUMMARY:
The purpose of this investigational study is to study the effects of Stimgenics Spinal Cord Stimulation (SGX-SCS) in subjects with chronic, intractable pain of the trunk with lower limb pain, including unilateral or bilateral pain associated with the following conditions: failed back surgery syndrome, intractable low back pain and leg pain.

DETAILED DESCRIPTION:
This is an open-label prospective, randomized, controlled, multi-center study comparing Stimgenics Spinal Cord Stimulation (SGX-SCS) programming approach to Standard SCS programming approach.

Subjects meeting study entrance criteria will be randomized in a 1:1 ratio to one of two study treatment groups:

* Test treatment group with SGX-SCS programming approach
* Control treatment group with Standard SCS programming approach

Data at follow-up visits will be compared between the two treatment groups, and in reference to baseline assessments collected at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be a candidate for SCS system (trial and implant) per labeled indication (back and leg pain)
2. Has an average back pain intensity ≥ 5.0 cm on the 10.0 cm Visual Analog Scale (VAS) at the time of enrollment with moderate to severe chronic leg pain
3. Be willing and capable of giving written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the subject's participation has been provided.
4. Be willing and capable of subjective evaluation, read and understand English-written questionnaires, and read, understand and sign the written inform consent in English.
5. Be 18 years of age or older at the time of enrollment
6. Be on a stable pain medication regime, as determined by the study investigator, for at least 30 days prior to enrolling in this study
7. Be willing to not increase pain medications from baseline through the 3-Month Visit
8. Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

1. Has a medical, anatomical, and/or psychosocial condition that is contraindicated for commercially available IntellisTM SCS systems as determined by the Investigator
2. Be concurrently participating in another clinical study
3. Has an existing active implanted device such as a pacemaker, another SCS unit, peripheral nerve stimulator, and/or drug delivery pump, etc.
4. Has pain in other area(s) and/or medical condition requiring the regular use of significant pain medications that could interfere with accurate pain reporting, study procedures, and/or confound evaluation of study endpoints, as determined by the Investigator
5. Has mechanical spine instability as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- StimGenics, Bloomington, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Arm | Control Arm
Started | 67 | 61
Completed | 67 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Arm | Control Arm | Total
Number analyzed (Participants) | 67 | 61 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.25 (12.16) | 60.66 (11.77) | 60.98 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 33 | 27 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 60 | 50 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Back Pain [Mean (Standard Deviation); unit: cm] — Visual Analog Score (0.0cm to 10.0cm line). Higher score represents more pain.
  cm | 7.25 (1.49) | 7.35 (1.26) | 7.3 (1.38)
Leg Pain [Mean (Standard Deviation); unit: cm] — Visual Analog Score (0.0cm to 10.0cm). Higher score represents more pain.
  cm | 6.2 (2.58) | 6.58 (2.06) | 6.38 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Individual Responders
Description: Percentage of Participants with a 50% decrease in back pain at 3 months compared to baseline. Pain rating will be measured on the 10 cm Visual Analog Scale (VAS). Change in back pain score will be used to determine individual responder (e.g., 50% reduction in VAS compared to Baseline VAS).
Time Frame: 3 months
Population: Intent to treat population (all subjects randomized)
Measure: Number (90% Confidence Interval); unit: percentage of responders
Groups:
- Control Arm: Subjects randomized to this arm will receive test treatment
  Standard SCS Programming Approach: Standard SCS Programming approach Using Intellis(TM) SCS system
Arm/Group | Test Arm | Control Arm
Number analyzed (Participants) | 67 | 61
percentage of responders | 80.9 [69.0 to 89.6] | 50.9 [39.1 to 62.6]

2. Secondary Outcome: Percentage of Individual Responders
Description: The percentage of Individual Responders (50% reduction in pain score rated on a Visual Analog Scale); Test for superiority
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Back Pain Score
Description: Comparison of change from Baseline in back pain score (using Visual Analog Scale 0.0-10.0cm) determined at the 3- and 6-month visit after device activation, between test and control in a statistical test of non-inferiority. This is calculated as: Change from Baseline in Back Pain VAS = 3-Month Visit Pain VAS - Baseline Pain VAS.
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: 6 Months Comparison of Back Pain Treatment Success
Description: Comparison of Back Pain Treatment Success (responder rate), measured as subjects with at least a 50% reduction in Back Pain Visual Analog Scale (VAS), evaluated at 6 months after device activation, between test and control
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Oswestry Disability Index (ODI)
Description: Oswestry Disability Index (ODI) evaluated at 3 months visit
Time Frame: 3 months
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events
Description: Frequency of treatment emergent adverse events
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events related to the study is collected.
Arm/Group | Test Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/67 | 2/61
Other Adverse Events (participants affected / at risk) | 0/67 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Arm (N=67) | Control Arm (N=61)
Implant Site Infection (Infections and infestations) | 0 | 1 (1)
Medical device site pain (General disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT03606187/Prot_SAP_000.pdf